CLINICAL TRIAL: NCT05127941
Title: Andexanet Alfa: Non-interventional Study in Stroke Units in Germany (DE)
Acronym: ASTRO-DE
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Hans Diener, Senior Professor of Clinical Neurosciences, University Hospital, Essen
Other Study IDs: ASTRO-DE
Record Dates: First submitted 2021-10-12; First posted 2021-11-19 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Intracranial Hemorrhages
Keywords: Intracranial bleeding; Andexanet-alfa; Rivaroxaban; Apixaban; Anticoagulation
MeSH Terms: conditions — Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient group: Patients under effective anticoagulation with rivaroxaban or apixaban and treated with andexanet alfa

SUMMARY:
The multicenter, prospective, observational, non-interventional study conducted in German Stroke Units is investigating patients with intracranial hemorrhage (ICH) under effective anticoagulation with rivaroxaban or apixaban.

The aim of the study is to analyze under routine conditions wether the volume increase of ICH under treatment with rivaroxaban and apixaban can be reduced with the antidote andexanet alfa. Thus, data of patients under effective treatment with rivaroxaban or apixaban and treated with andexanet alfa at baseline will be assessed at the time of onset of ICH, during the hospital stay and during a follow-up by telephone at 30 and 90 days after hospital discharge.

The main objective is defined as the change in size or volume of the hematoma by computed tomography (CT) or magnetic resonance imaging (MRI) in patients with ICH under effective treatment with rivaroxaban and apixaban, who are treated with andexanet alfa. Further objectives comprise evaluations concerning the functional status according to modified Rankin Scale (mRS), changes in the National Institutes of Health Stroke Scale (NIHSS), and occurrences of ICH or new intraventricular bleeding as well as mortality rates.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at enrollment
* Patients willing and able to provide written informed consent for data transmission. For patients who are not legally competent to sign this informed consent for data transmission exceptions/special cases are defined (details provided in the study protocol)
* Patients with primary intracranial hemorrhage as confirmed with CT or MRI.
* Patients under effective anticoagulation treatment with rivaroxaban or apixaban at the time of admission, according to the judgement of treating physician and determined using Point-of-care (PoC) anti-factor Xa (fXa) assays or laboratory-based anti-fXa measurement.
* Patients treated with andexanet alfa
* Signed informed consent as soon as possible after start of symptoms of initial ICH event, but before discharge

Exclusion Criteria:

* Start of symptoms of initial ICH event > 24 h before admission to hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with anticoagulating therapy with rivaroxaban or apixaban admitted with a clinically symptomatic ICH will be included in the study if they have been treated with andexanet alfa. A repeat CT or MRI between 12-72h after initial imaging to assess size and volume of bleeding corresponds to the standard treatment.
  The option to include patients under anticoagulating therapy edoxaban will be evaluated during the course of the study in case a marketing authorization of andexanet alfa for patients under edoxaban will be received.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Change in size (specified as ml or cm^3) of the intracranial bleeding evaluated by Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) | 12-72 hours after initial CT or MRI, further imaging in case of worsened health condition
  The primary endpoint is the change in size (specified as ml or cm^3) of the intracranial bleeding evaluated by first CT or MRI between 12-72 hours after initial CT or MRI; further imaging in case of worsened health condition

SECONDARY OUTCOMES:
Functional status according to modified Rankin Scale (mRS) | before ICH, at admission, at discharge, after 30 days, and after 90 days
  Functional status acc. to modified Rankin Scale (mRS) before ICH, at admission, at discharge, after 30 days, and after 90 days. The mRS ranges from grade 0 (no symptoms) to grade 6 (dead)
Mortality rate | after 7, 30 and 90 days und during hospital stay
  Mortality rate after 7, 30 and 90 days, and intra-hospital mortality rate
Rate of worsened health condition | At hospital admission and additionally at 24 hours and 72 hours after admission
  Rate of worsened health condition defined as change in NIHSS of ≥4 pts compared to initial NIHSS or worsening of NIHSS level of consciousness ≥1 point or increase of the volume of the intracranial bleeding or new intraventricular bleeding or death
Change in severity of stroke | 72 hours after admission
  Change in severity of stroke based on the National Institutes of Health Stroke Scale (NIHSS) 72 hours after admission
Assessment of effective anticoagulation at baseline | at baseline
  Assessment of effective anticoagulation at baseline using PoC anti-fXa assay, intra-hospital decision making for Andexanet alfa administration
Clinical course and outcomes of patients | Coagulation parameters will be recorded at hospital admission. Thrombotic events and re-bleeding will be recorded from the date of hospital admission until discharge. The average length of hospital stay is expected to be 10 days
  Hemostasis will be assessed by coagulation parameters (activated partial thrombin time (aPTT), thrombin time (TT), International Normalized Ratio (INR)) at admission, re-bleeding and thrombotic events (e.g. myocardial infarction, ischemic stroke, deep vein thrombosis) will be assessed by AE reporting performed from admission to hospital to discharge
Re-dosing and re-anticoagulation therapy | The assessement of re-dosing and re-anticoagulation therapy will take place from the date of hospital admission until the date of discharge. The average length of hospital stay is expected to be 10 days.
  Resumption of antithrombotic therapy in hospital (incl. type, start date and dose of anticoagulation therapy)
Health care resource utilization (including ICU length of stay) | Will be recorded during hospital stay until the date of discharge.The average length of hospital stay is expected to be 10 days.
  Data regarding ICU length of stay and on resource utilization (Intubated on arrival, Mechanical ventilation, ICH-evacuation surgery, External ventricular drainage, Intraventricular lysis, Osmotherapy)

OTHER OUTCOMES:
Safety endpoints | Will be recorded at hospital admission, at 24 and 72 hours after admission, at discharge. The average length of hospital stay is expected to be 10 days (depends on the severity of disease and cannot be specifically defined).
  Assessment of non-serious Adverse Events (AEs) and Serious Adverse Events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Hans Diener, Prof. Dr., Study Director — University Hospital, Essen
Locations (2):
- Germany (2):
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Tübingen, Tübingen